CLINICAL TRIAL: NCT05171842
Title: Safety and Efficacy of Endovascular Treatment in Patients With Spontaneous Isolated Superior Mesenteric Artery Dissection: a Multicenter, Prospective Single-arm Observational Study
Brief Title: Dissection of the Superior Mesenteric Artery
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Shandong Provincial Hospital (Other Government); Affiliated Hospital of Jiaxing University (Other); People's Hospital of Dangyang (Other); First People's Hospital of Hangzhou (Other); The First Affiliated Hospital of Anhui Medical University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: IIT20210045B
Record Dates: First submitted 2021-11-18; First posted 2021-12-29 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Dissection of the Superior Mesenteric Artery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Observe the prognosis after stent implantation — Observe the prognosis of patients after undergoing specific operations. Specific surgery: Use femoral artery or brachial artery to implant bare stent (stent with diameter ≤7mm is suggested to use thin-wall stent, stents with >7mm are not restricted) to restore the blood flow of the true lumen superior mesenteric artery. If the false cavity is large, it can be combined with a spring coil to assist embolization. Anticoagulant therapy should be performed for at least 1 day after surgery. Anticoagulant drugs are not restricted. After discharge from the hospital, the dual anti-platelet drugs should be taken for 3 months, and a single anti-platelet drug should be maintained for at least 1 year.

SUMMARY:
This study aims to evaluate the prognosis of patients with spontaneous solitary dissection of superior mesenteric artery (SIDSMA) who have been treated with stents.

DETAILED DESCRIPTION:
This study is an observational study. The subject's treatment plan needs to be expected to meet the following conditions: the corresponding surgery has been completed: the femoral artery or brachial artery approach is implanted into the true lumen of the SMA bare stent (the part with a diameter ≤ 7mm is suggested to use thin-wall stent, and the part with a diameter> 7mm It is not limited to using stents (brands) to restore the real lumen blood flow of the superior mesenteric artery. If the false cavity is large, it can be combined with a spring coil to assist embolization. Anticoagulation therapy for at least 1 day after surgery. Anticoagulation drugs are not limited to use. After discharge, the dual-antiplatelet drugs for at least 3 months, and single antiplatelet should be maintained for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Superior mesenteric artery dissection with obvious abdominal symptoms within 1 month of onset

  * CTA/DSA diagnosed as spontaneous superior mesenteric artery dissection; ③ CTA/DSA diagnosed as a solitary superior mesenteric artery dissection; ④ Sign the informed consent form and be willing to accept follow-up observation;

Exclusion Criteria:

1. Those suffering from mental illness or subjectively unable to cooperate;
2. Patients with asymptomatic spontaneous solitary superior mesenteric artery dissection or only superior mesenteric artery intermural hematoma;
3. Patients with signs of peritonitis (tenderness, rebound pain, flat abdomen) and suggest severe intestinal ischemia;
4. Patients with strangulated intestinal obstruction;
5. Other patients who plan to undergo open surgery;
6. Women who are breastfeeding or pregnant, or women or men who have recent birth plans;
7. Life expectancy <2 years;
8. Patients who are currently participating in other interventional drug or device research, or have been enrolled in this research;
9. Patients with renal failure or chronic kidney disease have MDRD GFR ≤ 30ml/min/1.73 m2 (or serum creatinine ≥2.5 mg/dL within 30 days before surgery, or receive dialysis treatment);
10. Diagnose active systemic infection or uncontrolled coagulation dysfunction within 14 days before operation;
11. History of previous superior mesenteric artery surgery;
12. Failure to take medications as required by the protocol, or allergy to antiplatelet drugs (aspirin or clopidogrel), low molecular weight heparin, vasodilators or contrast agents, so that the preoperative and postoperative medication requirements cannot be fully complied with
13. Combined with systemic diseases that cannot be controlled by the current medical level (such as severe heart function, lung function or liver function abnormalities, patients with advanced tumors, patients with cachexia, patients with severe coronary heart disease that cannot be relieved, abnormal blood coagulation caused by genetic diseases, etc.)
14. Cerebral hemorrhage, symptomatic stroke, myocardial infarction, gastrointestinal hemorrhage in the past 6 months or the patient is under 18 years of age or the patient refuses to participate in the study
15. Does not meet the expected intraoperative and postoperative treatment plan
16. The diameter of the true lumen in the anchoring area of the SMA distal stent is less than 3mm

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: SIDSMA patients receiving stent therapy
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Re-intervention rate at 12 months after endovascular treatment | 12months
  Including surgery related to this disease (including surgical intervention at the puncture point) and symptom recurrence requires more than 3 days of conservative treatment

SECONDARY OUTCOMES:
Disease-related mortality at 1, 6, and 12 months after surgery | 1/6/12months
  Disease-related mortality at 1, 6, and 12 months after surgery
Stent patency rate at 1, 6, and 12 months after surgery | 1/6/12months
  Stent patency rate at 1, 6, and 12 months after surgery
Dissection shape at 1, 6, and 12 months after surgery | 1/6/12months
  Dissection shape at 1, 6, and 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hongkun zhang, Study Chair — First Affiliated Hospital of Zhejiang University
Locations (1):
- First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Qiu C, He Y, Li D, Shang T, Wang X, Wu Z, Zhang H. Mid-Term Results of Endovascular Treatment for Spontaneous Isolated Dissection of the Superior Mesenteric Artery. Eur J Vasc Endovasc Surg. 2019 Jul;58(1):88-95. doi: 10.1016/j.ejvs.2018.11.013. Epub 2019 May 31. PMID 31160187
- [Background] Wang B, Pan J, Xu Y, Qiu X, Ding Z, Li D, Zhang H, Qiu C, Wu Z. Long-term Outcomes of Endovascular Versus Medical Treatment for Isolated Superior Mesenteric Artery Dissection: A 10-Year Retrospective Study. Cardiovasc Intervent Radiol. 2025 May;48(5):593-602. doi: 10.1007/s00270-025-03985-0. Epub 2025 Feb 26. PMID 40011282
- [Background] Qiu C, Wu Z, He Y, Tian L, Zhu Q, Shang T, Zhang H, Li D. Endovascular therapy versus medical treatment for spontaneous isolated dissection of the superior mesenteric artery. Cochrane Database Syst Rev. 2022 Sep 8;9(9):CD014703. doi: 10.1002/14651858.CD014703.pub2. PMID 36074662